CLINICAL TRIAL: NCT04030559
Title: Phase II Trial of PARP Inhibitor Niraparib for Men With High Risk Prostate Cancer and DNA Damage Response Defects
Brief Title: Niraparib Before Surgery in Treating Patients With High Risk Localized Prostate Cancer and DNA Damage Response Defects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marc Dall'Era, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Janssen, LP (Industry)
Responsible Party: Sponsor-Investigator, Marc Dall'Era, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1412676; NCI-2019-04365 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#279 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: ATM Gene Mutation; BRCA1 Gene Mutation; BRCA2 Gene Mutation; BRIP1 Gene Mutation; CDK12 Gene Mutation; CHEK1 Gene Mutation; CHEK2 Gene Mutation; DNA Damage Response Gene Mutation; DNA Repair Gene Mutation; FANCA Gene Mutation; FANCD2 Gene Mutation; FANCL Gene Mutation; GEN1 Gene Mutation; NBN Gene Mutation; Prostate Carcinoma; RAD51 Gene Mutation; RAD51C Gene Mutation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (niraparib) (Experimental): Patients receive niraparib PO QD on days 1-28. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Following completion of treatment, patients then undergo standard of care surgery.
  Interventions: Drug: Niraparib; Drug: Niraparib Tosylate Monohydrate; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Niraparib — Given PO
  Other Names: MK-4827; MK4827
Drug: Niraparib Tosylate Monohydrate — Given PO
  Other Names: Zejula
Procedure: Radical Prostatectomy — Undergo standard of care surgery
  Other Names: Prostatovesiculectomy

SUMMARY:
This phase II trial studies how well niraparib, when given before surgery, works in treating patients with high risk prostate cancer that has not spread to other parts of the body (localized) and alterations in deoxyribonucleic acid (DNA) repair pathways. Niraparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the impact of neoadjuvant niraparib tosylate monohydrate (niraparib) therapy prior to radical prostatectomy (RP) on pathologic tumor stage, frequency of lymph node metastases and positive margin rates for patients undergoing radical prostatectomy for high-risk, clinically localized prostate cancer with alterations in DNA repair pathways.

SECONDARY OBJECTIVE:

I. To assess 5-year biochemical recurrence in subjects with high-risk prostate cancer and DNA-damage response defects after prostatectomy.

OUTLINE:

Patients receive niraparib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Following completion of treatment, patients then undergo standard of care surgery.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 2 years, and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and other protocol requirements
* Patients must have histologically or cytologically confirmed prostate cancer that is clinically localized as defined by negative cross-section imaging and/or bone scan, and classified as high or very high risk per National Comprehensive Cancer Network (NCCN) guideline
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1
* Life expectancy >= 10 years
* Men who have selected radical prostatectomy as the primary treatment for their prostate cancer
* Prostate cancer tumors with alterations in key DNA repair genes. This will include at least one alteration in a gene involved in DNA repair primarily through the homologous recombination pathway including BRCA1/2, ATM, CHEK1/2 FANCA, FANCD2, FANCL, GEN1, NBN, PALB2, RAD51, RAD51c, and BRIP1. Mutations will be selected that are known or likely pathogenic. Mean allele frequencies will be assessed to estimate mono versus biallelic loss of function. Patients with biallelic deletions or mutations will be prioritized for inclusion to make up at least 30% of the enrollment (i.e., 10 patients) to gauge response in this group over monoallelic loss. Final inclusion will be determined by the principal investigator
* Must be able to swallow whole capsules
* To avoid risk of drug exposure through the ejaculate, male subjects (even if they have undergone a successful vasectomy) must agree while on study therapy (including during dose interruptions) and for 3 months following the last dose of study drug to:

  * Use a condom during sexual activity or practice complete sexual abstinence
  * Not donate sperm
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (obtained =< 14 days of the first study treatment)
* Platelet count >= 100 x 10^9/L (obtained =< 14 days of the first study treatment)
* Hemoglobin >= 9 g/dL (may have been transfused) (obtained =< 14 days of the first study treatment)
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN) range (obtained =< 14 days of the first study treatment)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels =< 2.5 x ULN or AST and ALT levels =< 5 x ULN (for subjects with documented metastatic disease to the liver) (obtained =< 14 days of the first study treatment)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (for patients on anticoagulation they must be receiving a stable dose for at least 1 week prior to randomization) (obtained =< 14 days of the first study treatment)
* Creatinine clearance > 30 mL/min by Cockcroft-Gault formula (or local institutional standard method) (obtained =< 14 days of the first study treatment)

Exclusion Criteria:

* Any condition that would prohibit the understanding or rendering of informed consent
* Prior treatment for prostate cancer
* Prior treatment with a PARP inhibitor
* Prior treatment with androgen deprivation therapy (luteinizing hormone-releasing hormone [LHRH] agonist/antagonist), antiandrogen (e.g., bicalutamide, nilutamide, enzalutamide, apalutamide), or androgen synthesis inhibitor (e.g., abiraterone, orteronel)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Uncontrolled concomitant disease that in the opinion of the investigator would interfere with the patient's safety or compliance on trial
* Severe infection that in the opinion of the investigator would interfere with the patient's safety or compliance on trial within 4 weeks prior to enrollment
* Known allergies, hypersensitivity, or intolerance to niraparib or its excipients (refer to investigator's brochure)
* Known disorder affecting gastrointestinal absorption
* Corrected QT interval by the Fridericia correction formula (QTcF) on the screening electrocardiography (ECG) > 450 msec
* Receiving concomitant medications that prolong QTc and are unable to discontinue use while receiving study drug
* History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
* Known human immunodeficiency virus (HIV) positive subjects with 1 or more of the following:

  * Not receiving antiretroviral therapy
  * A change in antiretroviral therapy within 6 months of the start of screening (except if, after consultation with the sponsor, a change is made to avoid a potential drug-drug interaction with the study drug)
  * Receiving antiretroviral therapy that may interfere with the study drug (consult the principal investigator [PI] for review of medication prior to enrollment)
  * CD4 count < 350 at screening
  * An acquired immunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate (pRR) | At the time of radical prostatectomy procedure
  The study will assess the impact of neoadjuvant niraparib therapy prior to radical prostatectomy (RP) on pathologic tumor stage, frequency of lymph node metastases and positive margin rates for patients undergoing radical prostatectomy for high-risk, clinically localized prostate cancer with alterations in deoxyribonucleic acid (DNA) repair pathways. Pathologic complete response (PCR) defined as no tumor identified on hematoxylin and eosin (H&E) stained sections will be assessed; minimal residual disease (MRD) will be defined as tumor clusters limited to < 5 mm and confined to prostate gland.
  Exact 95% confidence intervals for pRR and other binary outcomes, adjusted for the two-stage design, will be calculated as described by Koyama and Chen. Response rates will be compared between patients with biallelic and monoallelic loss using Fisher's Exact Test.

SECONDARY OUTCOMES:
Biochemical prostate specific antigen (PSA) progression free survival | Up to 5 years
  Median biochemical progression free survival (bPFS) and quartiles (when reached) will be calculated from Kaplan-Meier estimates, and 95% confidence intervals will be calculated using Greenwood's formula.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dall'Era, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- [Derived] Montgomery B, Mostaghel EA. Neoadjuvant Therapy Prior to Prostatectomy: Is the Glass Half Full? Eur Urol. 2023 Jun;83(6):519-520. doi: 10.1016/j.eururo.2023.01.021. Epub 2023 Jan 27. No abstract available. PMID 36710203
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-experimental-medicine-niraparib-for-men-with-high-risk-prostate-cancer-713066/